CLINICAL TRIAL: NCT02602210
Title: Supplemental Corticosteroids in Cirrhotic Hypotensive Patients With Suspicion of Sepsis
Acronym: SCOTCH;
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low inclusion rate
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCOTCH-SCotCHIS in the UK
Record Dates: First submitted 2015-09-22; First posted 2015-11-11 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Liver Cirrhosis
Keywords: cirrhosis; liver; corticosteroids; hypotension; sepsis; cortisol
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Hypotension; Sepsis | interventions — Hydrocortisone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Active Comparator): Group A: treated with intravenous hydrocortisone in addition to standard therapy (= treatment group)
  Interventions: Drug: Hydrocortisone
- group B (Placebo Comparator): Group B: IV treatment with NaCL 0.9% in addition to standard therapy (= placebo group)
  Interventions: Drug: NaCL 0.9%

INTERVENTIONS:
Drug: Hydrocortisone — IV bolus of 100 mg hydrocortisone in 50ml NaCl 0.9% (sodium chloride); followed by continuous IV infusion of 200 mg hydrocortisone in 50 ml NaCl 0.9% at a rate of 2 ml/h until the start of day 4.Reduction of infusion rate with 0.5 ml/h/day.
  Other Names: solucortef
  Arms: group A
Drug: NaCL 0.9% — IV bolus of 50 ml NaCL 0.9%; followed by continuous IV infusion of NaCL 0.9%
  Other Names: sodium chloride
  Arms: group B

SUMMARY:
The main goal of the study is to investigate the clinical relevance, efficacy and safety of treating hypotensive cirrhotic patients with suspicion of sepsis and on vasopressors with low-dose hydrocortisone in order to reverse hemodynamic instability and organ failure and to decrease mortality.

DETAILED DESCRIPTION:
Ample evidence suggests that a significant number of patients (52-77%) with chronic liver disease develop adrenal insufficiency in case of concomitant sepsis. This condition impairs hemodynamic integrity and probably worsens often encountered multiorgan failure. Different groups suggested that treating those patients with corticosteroids gives a faster reversal of hemodynamic instability and even lowers mortality compared to historical controls. However, most of the published data are retrospective and comprise small groups of patients. These data raise the possibility that corticosteroids at stress doses may be beneficial in hypotensive cirrhotics admitted to the ICU but as yet this has not been subjected to a large-scale multicentre randomized controlled clinical trial.

The study will be a double-blind, randomized, placebo-controlled, multicenter trial, involving tertiary intensive care units with expertise in management of patients with decompensated cirrhosis. Patients who satisfy inclusion criteria and do not present any of the exclusion criteria at ICU admission will be randomized into two groups:

* Group A: treated with intravenous hydrocortisone in addition to standard therapy (= treatment group)
* Group B: placebo (NaCl 0.9%) treatment in addition to standard treatment (= placebo group)

If, after adequate fluid resuscitation, patients are still on norepinephrine at a dose of at least 0,1 mcg/kg/min for at least 4 hours, the patient can be randomized. Study drug can be started immediately after randomization but no later than 24 h after initiation of norepinephrine. Patients will receive an intravenous bolus of 50 ml of normal saline (placebo) or an intravenous bolus of 50 ml of normal saline containing 100 mg of hydrocortisone (double-blind) that will be followed by a continuous intravenous infusion of the study drug (hydrocortisone) or placebo. Treatment with study drug (hydrocortisone or placebo) at initial rate will be maintained until the start of day 4 and gradually discontinued (reduction of infusion rate with 0.5 ml/h/d) when 1) patients do not require vasoactive drugs anymore to maintain MAP(mean arterial pressure) > 60 mmHg or > 65 mmHg if associated with signs of hypoperfusion in spite of ongoing adequate fluid resuscitation or 2) in any case after a 7-day treatment period.

Investigators, treating physicians, nurses and patients will be blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* All patients with known or recently diagnosed cirrhosis who

  1. are admitted to the ICU because of persistent hypotension or
  2. develop persistent hypotension while admitted to the ICU,

secondary to proven or suspected infection, in both cases despite adequate fluid resuscitation and with persistent need for low-dose norepinephrine to maintain a mean arterial blood pressure > 60 mmHg or > 65 mmHg if accompanied by signs of hypoperfusion, are eligible for study entry. The diagnosis of cirrhosis is preferably made by histology or based on imaging and laboratory findings.

Exclusion Criteria:

* Age < 18 or ≥ 80 years
* Patients receiving any vasopressor medication for more than 24 h prior to administration of study drug. Terlipressin initiated for treatment of hepatorenal syndrome or variceal bleeding is allowed
* Patients with known hypoadrenalism
* Active GI bleeding (unless controlled for >72 hours) or hemorrhagic shock.
* Cardiogenic shock or severe cardiac dysfunction (CI <2 l/min/ m2)
* Active uncontrolled hepatitis B infection
* HIV infection
* Evidence of current malignancy (except hepatocellular carcinoma within transplant criteria or non-melanocytic skin cancer)
* Therapy with any corticosteroid (oral or intravenous) in the last 3 months
* Patients who received etomidate within the past 3 days
* Severe acute alcoholic hepatitis (biopsy proven)
* Chronic hemodialysis
* Severe chronic heart disease (NYHA class III or IV)
* Severe chronic obstructive pulmonary disease (GOLD III or IV)
* Severe psychiatric disorder
* Child-Pugh score C14 -15
* SOFA score > 16 points at inclusion
* Pregnant or breastfeeding women
* Contraindications for systemic steroids
* Refusal to consent
* Patients who cannot provide prior informed consent and when there is documented evidence that the patient has no legal surrogate decision maker and it appears unlikely that the patient will regain consciousness or sufficient ability to provide delayed informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Patient survival at 28 days analysed from the day of randomisation | 28days
  survival status

SECONDARY OUTCOMES:
patient survival at 90 days analysed from the day of randomization | 90 days
  survival status
ICU and hospital mortality | from the date of randomisation until ICU discharge or hospital mortality, whichever came first, up to day 90
  mortality
reversal of shock | up to day 90
  time in days from start of placebo or active medication to resolution of shock as defined as cessation of continuous vasopressor medication (for > 24 hours)
reversal of organ failures | up to 90 days
  measured with SOFA-score and CLIF (Chronic Liver Failure Consortium)-SOFA score
vasopressor doses | up to 90 days
  administration of vasopressor
vasopressor-free days | up to 90 days
  days without vasopression
mechanical ventilation-free days | up to 90 days
  days without mechanical ventilation
need for and duration of renal replacement therapy | up to 90 days
  days of renal replacement therapy
ICU and hospital length-of-stay | up to 90 days
  days of ICU stay , days of hospital stay
acquirement of new infections | up to 90 days
  bacterial and/or fungal: defined according to CDC (Centers for Diseases Control) criteria (pneumonia, bacteremia, spontaneous bacterial peritonitis, catheter-related bloodstream infections, skin infections and others)
shock relapse | during tapering period until 3 days after end of study drug
  defined as hypotension recurrence during the tapering period or within 3 days of total discontinuation of study drug
clinically important bleeding | up to 90 days
  defined as new melena, new haematemesis or unexplained fall in haemoglobin > 2g/dl (not related to volume expansion). The presence of 'coffee ground' aspirate from nasogastric aspirate will not be considered active GI bleeding.
glycemic control | during ICU stay, up to 10 days
  measured as units of insulin required to attain glycemic levels between 80 - 140 mg/dl
episode of hyper- (> 180 mg/dl) or hypoglycemia (< 60 mg/dl) | during study treatment period, up to 10 days
  number of episodes of hypo- hyperglycemia
new shock episode | during study treatment period, up to 13 days
  hypotension recurrence with need for vasopressor therapy after 3 days of total discontinuation of study drug
impact of coagulopathy | during ICU stay up to 10 days
  assessed by disseminated intravascular coagulopathy (DIC)-score
incidence of ICU-acquired weakness | during ICU stay, up to 90 days
  occurrence of IC acquired weakness

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Meersseman, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Alexander Wilmer, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Javier Fernandez, MD,PhD, Principal Investigator — Hosp Clinic, Barcelona, Spain
Locations (10):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams Brabant, Belgium
- Institute for Clinical and Experimental Medicine, Prague, Czechia
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- San Giovanni Battista Hospital, Turin, Italy
- Spain (3):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
- United Kingdom (2):
  - King's College Hospital, London
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Meersseman P, Hernandez-Tejero M, Diaz JM, Wauters J, Hermans G, Aziz F, Ceunen H, Prado V, Langouche L, Arteaga M, Acevedo J, Lleixa M, Zapatero J, Toapanta D, Arroyo V, Wilmer A, Fernandez J. Low-Dose Hydrocortisone in Cirrhotic Patients With Septic Shock: A Double-Blind Randomised Placebo-Controlled Trial. Liver Int. 2025 Sep;45(9):e70257. doi: 10.1111/liv.70257. PMID 40757786